CLINICAL TRIAL: NCT00794352
Title: Comprehensive Multimodal Analysis of Patients With Neuroimmunological Diseases of the CNS
Brief Title: Comprehensive Multimodal Analysis of Neuroimmunological Diseases of the Central Nervous System
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090032; 09-I-0032
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-08

CONDITIONS: Central Nervous System Disease; Multiple Sclerosis
Keywords: Inflammation; Multiple Sclerosis; Neuroimmunology; Immune Disorder; Neuroimaging; Natural History; Central Nervous System Disease; Healthy Volunteers; HV
MeSH Terms: conditions — Central Nervous System Diseases; Multiple Sclerosis; Inflammation; Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: Healthy patients with NO inflammatory and/or demyelinating/dysmyelinating diseases of the CN
- Patient Cohort: Patients who present with CNS white matter injury (including inflammatory and/or demyelinating/dysmyelinating diseases of the CNS)

SUMMARY:
Inflammatory or degenerative diseases of the brain and spinal cord, such as multiple sclerosis, may be related to problems with an individual s immune system. However, more information is needed on the ways in which the cells of the immune system interact with the central nervous system (CNS). This study will compare tests performed on both healthy volunteers and individuals who have signs or symptoms of immune-related damage to their CNS.

This study will include two groups of subjects at least 12 years old. Subjects will either have symptoms of immune-related CNS damage, or will be healthy volunteers selected for comparison purposes.

Study participants will visit the NIH Clinical Center on an outpatient basis for an initial evaluation visit. During the visit, patients will provide a comprehensive medical history and undergo a neurological examination, and will provide blood samples for research purposes. The healthy volunteers will be asked to schedule a return visit for a magnetic resonance imaging (MRI) procedure, and may be asked to undergo other tests requested by the study researchers on an as-needed basis. The group of patients with symptoms of immune-related CNS damage will be asked to undergo a series of tests, including the following:

* MRI procedures, with a minimum of three brain MRIs and one spinal cord MRI taken approximately 4 weeks apart
* A diagnostic lumbar puncture, performed on an outpatient basis
* Tests of brain and vision activity
* Additional blood and tissue samples

Patients with symptoms of immune-related CNS damage may be offered the opportunity to participate in additional followup tests with NIH researchers.

DETAILED DESCRIPTION:
OBJECTIVE

The goal of this study is to define the pathophysiological mechanisms underlying the development of disability in immune-mediated disorders of the central nervous system (CNS) and to distinguish these from beneficial responses of the human immune system to CNS injury.

The protocol serves as a screening tool for Neuroimmunological Diseases Section (NDS) of the National Institute of Allergy and Infectious Diseases (NIAID) clinical trials and enables development of clinically-useful tools such as diagnostic tests and new, sensitive scales of neurological disability, disease severity and CNS tissue destruction.

This protocol also serves as a repository to enable prospective institutional review board (IRB) review of research using human samples and data collected under other NDS protocols.

STUDY POPULATION

Patients with evidence, or suspicion of immune-mediated CNS injury. Healthy volunteers (HV) are included as controls for immunological and imaging biomarkers and to obtain normative data for development of new clinical scales and smartphone apps.

DESIGN

Collection of multimodal data (standardized clinical/functional, neuroimaging and molecular/immunological data) during the diagnostic work-up of patients with varied disorders of the CNS in which immune-mediated processes are expected to play a pathophysiological role.

For the patient cohort, a comprehensive evaluation establishes a definitive diagnosis or confirms diagnosis and subtype of multiple sclerosis (MS) as a pre-requisite for enrollment into NDS clinical trials. Adult patients have a mandatory follow-up visit approximately 1-2 years from protocol enrollment. Depending on the diagnosis and clinical/research needs, patients may be offered additional follow-up visits. The maximum frequency of the follow-up visits and research samples to be collected is specified to ensure patient safety. Patients age 12-17 years are included in the patient cohort to establish a definitive diagnosis, or to provide non-standard assays to help with diagnostic and therapeutic decisions as part of extraordinary clinical care.

The HV provide sex and age-matched (to adult patients) normative values.

A "telemedicine" patient sub-cohort enrolls patients who cannot (for any reason, but usually advanced disability) come to NIH for in-person evaluation. From these telemedicine patients, we will estimate neurological disability by Combinatorial MRI Scale (COMRIS) models derived from outside brain and spinal cord MRIs, and by NeuFun-TS smartphone application. Telemedicine patients will contribute capillary blood from at-home collection kits for research applications. Telemedicine patients with confirmed diagnosis of neuroimmunological disorder may be referred to NIAID Centralized Sequencing protocol (17-I-0122) for genetic testing.

A "sample processing only" patient subcohort enrolls patients from whom only biological samples and data collected by outside clinicians are processed and evaluated to provide non-standard assays.

A collaboration was in place until December 26, 2022, with the U.S. Food & Drug Administration that included collection of clinical and normative data for diagnostic and research purposes. The FDA Principal Investigator Dr. Wenyu Sun will assist with the needs of the protocol by performing minimal protocol related procedures. Such procedures are discussed throughout Study Design and Methods.

OUTCOME MEASURES

Clinical, MRI, and immunological outcomes are outlined in this section. However, no pre-defined research questions will be addressed other than to establish the diagnosis, determine the level of disability, provide prognostic information, and monitor the natural history.

ELIGIBILITY:
* PATIENT INCLUSION CRITERIA (for in-person and telemedicine sub-cohorts):

Presentation with a clinical syndrome consistent with immune-mediated CNS disorder and/or

Neuroimaging evidence of inflammatory and/or demyelinating/dysmyelinating CNS disease

At least 12 years old at the time of enrollment

Willing to share medical records (including past MRI results) with the study team.

Adults: Able to give informed consent on their own or via a Legally Authorized Representative (LAR) or Durable Power of Attorney (DPA); or Minors: parent or legal guardian able to give consent, with child willing to give assent, if reasonable based on their age and assent capacity

For in-person sub-cohort: Able to undergo the required procedures, including LP, MRI and clinical/functional evaluations

PATIENT EXCLUSION CRITERIA (for in-person and telemedicine sub-cohorts):

Significant medical condition that would make participation in research part of evaluation impossible or risky

For in-person sub-cohort: Medical contraindications for MRI (i.e. any non-organic implant or other device such as a cardiac pacemaker or infusion pump or other metallic implants, objects or body piercings that cannot be removed)

Unwilling to consent for collection of biological samples or their cryopreservation

PATIENT INCLUSION CRITERIA for processing of collected biological samples:

Presentation with a clinical syndrome consistent with immune-mediated CNS disorder and/or

Neuroimaging evidence of inflammatory and/or demyelinating/ dysmyelinating CNS disease

Ability to obtain either direct or surrogate informed consent for sample processing and storage

Aged 0+ years

HEALTHY VOLUNTEER (in person) INCLUSION CRITERIA:

At least 18 years old at the time of enrollment

Vital signs are found within normal range at the time of the screening visit

Able to give informed consent

Able and willing to undergo related research procedures, such as blood draw, LP

HEALTHY VOLUNTEER (in person) EXCLUSION CRITERIA:

Systemic inflammatory disorder, or inflammatory or non-inflammatory neurological diseases

Previous or current history of alcohol and substance abuse

Medical contraindications for MRI (i.e. any non-organic implant or other device such as a cardiac pacemaker or infusion pump or other metallic implants, objects or body piercings that cannot be removed)

Medical contraindication for LP

Psychological contraindications for MRI (i.e. claustrophobia). This will be assessed at the time the medical history is collected

Pregnancy or current breastfeeding

Any contraindications to having study procedures done

History of auditory disorder (i.e. hearing impairment, known impaired acoustic reflex, tinnitus)

HEALTHY VOLUNTEER SUB-STUDY TO OBTAIN NORMATIVE DATA FOR THE SMARTPHONE APPS:

Because this sub-study collects no personal identifiable information (PII), there are no inclusion/exclusion criteria. Participating subjects are self-declared as not having any neurological deficit, which would be the same population that would provide normative data if the apps were freely available via App store.

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with evidence, or suspicion of immune-mediated CNS injury will be enrolled. In addition, healthy volunteers will be included as controls for immunological and imaging biomarkers and to obtain normative data for development of new clinical scales and smartphone apps.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2008-10-01 (Actual)

PRIMARY OUTCOMES:
Disease progression as assessed by clinical and MRI criteria. | 1-2 years
  1. Sustained (i.e. > 3 months) progression of disability as measured by => 0.5 CombiWISE points or 2. Development of new/clearly enlarged distinct lesions on T2WI
Definite diagnosis of MS or another disorder. | 12 weeks
  To identify MS-specific markers, biomarkers from peripheral blood and CSF will be compared between patients who fulfilled diagnostic criteria for MS versus those who were found to have alternative diagnoses.

SECONDARY OUTCOMES:
MRI measures of lesion load and CNS tissue destruction | within 1 week of first NDS visit
  for initial evaluation
Immunological biomarkers | Within 1 week of initial CSF
  for initial evaluation
Clinical measures of disability | within 1 week of follow-up visit
  for longitudinal evaluation
Changes in MRI measure of lesion load and CNS tissue destruction from baseline | within 1 week of follow-up visit
  for longitudinal evaluation
Changes in clinical measures of disability from baseline | within 1 week of initial NDS MRI
  for initial evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Bielekova, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim Y, Varosanec M, Kosa P, Bielekova B. Confounder-adjusted MRI-based predictors of multiple sclerosis disability. Front Radiol. 2022 Sep 13;2:971157. doi: 10.3389/fradi.2022.971157. eCollection 2022. PMID 37492673
- [Derived] Kosa P, Masvekar R, Komori M, Phillips J, Ramesh V, Varosanec M, Sandford M, Bielekova B. Enhancing the clinical value of serum neurofilament light chain measurement. JCI Insight. 2022 Aug 8;7(15):e161415. doi: 10.1172/jci.insight.161415. PMID 35737460
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-I-0032.html